CLINICAL TRIAL: NCT05626335
Title: Does Double (Fixed and Removable Orthodontic Retention) With Regular Monitoring Prevent Undesired Tooth Movement?
Brief Title: Does Double With Regular Monitoring Prevent Undesired Tooth Movement?
Status: Completed | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Collaborators: 3Shape Poland Sp.z.o.o. (Unknown); Koszalin University of Technology (Unknown)
Responsible Party: Sponsor
Other Study IDs: KB-0012/74/10/2020/Z
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-10

CONDITIONS: Malocclusion
Keywords: retention; stability; orthodontic treatment; 3D analysis; intraoral scan
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: From all the patients meeting the inclusion criteria every third patients was randomly chosen and invited to participate in the study. Written informed consent was obtained from every participant. Thus 100 patients have agreed to participate. All fixed retainers (stainless steel braided rectangular wire) were bonded in both arches by the same experienced clinician, who subsequently made impression for thermally formed splints and delivered them on the day of debonding. The effect of each of the procedures was verified by two independent experienced clinicians. On the day of debonding, directly following retainer bonding, intraoral scans were performed (T0). The patients were invited for repeating the scans after 1 (T1), 3 (T2) and 6 months (T3). The displacements were assessed by superimposition of the scans. The patients were recommended to wear removable retainers 22h/day. They were instructed to immediately report a failure and to apply immediately to the office in case of failure.
  Interventions: Diagnostic Test: Intraoral scan

INTERVENTIONS:
Diagnostic Test: Intraoral scan — On the day of debonding, directly following retainer bonding, intraoral scans were performed (T0), using 3Shape Trios 4 (3Shape, Copenhagen, Denmark). The scans were repeated after a month. The patients were invited for repeating the scans after 1 (T1), 3 (T2) and 6 months (T3).

SUMMARY:
The goal of observational study is to learn about the stability of orthodontic treatment results in orthodontic patients during retention phase of treatment.

DETAILED DESCRIPTION:
The aim of the present study was to three-dimensionally analyze tooth movement in retention phase of treatment and wherever double effectively retention prevents it.

ELIGIBILITY:
Inclusion Criteria:

* Non-extraction treatment
* No hypodontia
* Normal occlusion after treatment (Class I occlusion), perfect alignment
* Normal overjet and overbite
* Double retention including fixed retainer bonded from canine to canine in both dental arches and thermally formed removable splint

Exclusion Criteria:

* Fixed orthodontic treatment in one dental arch
* Extraction cases
* Patient treated with orthognathic surgery
* Imperfect treatment result due to treatment cessation on patients demand or health issues
* Craniofacial disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group comprised 300 patients adult patients (age 18 to 41) who have completed fixed orthodontic treatment between (1st January 2021 - 9th September 2022).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Tooth displacement in mm | One month after debonding
  Measurement obtained by comparing superimposed scans
Tooth displacement in mm | Three months after debonding
  Measurement obtained by comparing superimposed scans
Tooth displacement in mm | Six months after debonding
  Measurement obtained by comparing superimposed scans

SECONDARY OUTCOMES:
Failure rate | Six months of observation
  Registration wherever the retention failure occured
Compliance rate | Six months of observation
  Registration of patients attending to scheduled visits

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Interdisciplinary Dentistry, Pomeranian Medical Univeristy in Szczecin, Szczecin, West Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No